CLINICAL TRIAL: NCT05613478
Title: Camrelizumab Combined With Apatinib Mesylate and TACE in the Perioperative Treatment of Hepatocellular Carcinoma: a Randomized, Open-label, Parallel, Multicenter Trial
Brief Title: Camrelizumab Combined With Apatinib Mesylate and TACE in the Perioperative Treatment of Hepatocellular Carcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Xuehao Wang, professor, The First Affiliated Hospital with Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022-SR-558
Record Dates: First submitted 2022-11-06; First posted 2022-11-14 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Hepatocellular Carcinoma; Immunotherapy; Preoperative
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — camrelizumab; apatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Preoperative TACE treatment → preoperative camrelizumab combined with apatinib mesylate (q2w, 2 cycles) → radical surgery → sequential camrelizumab and apatinib mesylate (q3w, at least 6 cycles)
  Interventions: Drug: Camrelizumab; Drug: Apatinib Mesylate; Procedure: Radical surgery; Procedure: Preoperative TACE treatment
- Control group (Active Comparator): Radical surgery → sequential camrelizumab and apatinib mesylate (q3w, at least 6 cycles)
  Interventions: Procedure: Radical surgery; Drug: Camrelizumab; Drug: Apatinib Mesylate

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab is administered at 200mg, q2w (2cycles) before radical surgery and 200mg, q3w (at least 6 cycles) after radical surgery
  Arms: Experimental group
Drug: Apatinib Mesylate — Apatinib Mesylate is administered at 250mg, qd (2 cycles) before radical surgery and 250mg, qd (at least 6 cycles) after radical surgery
  Arms: Experimental group
Procedure: Radical surgery — Radical surgery
Procedure: Preoperative TACE treatment — TACE treatment before preoperative camrelizumab combined with apatinib mesylate
  Arms: Experimental group
Drug: Camrelizumab — Camrelizumab is administered at 200mg, q3w (at least 6 cycles) after radical surgery
  Arms: Control group
Drug: Apatinib Mesylate — Apatinib Mesylate is administered at 250mg, qd (at least 6 cycles) after radical surgery
  Arms: Control group

SUMMARY:
Hepatocellular carcinoma (HCC) is the most common primary liver cancer. Hepatectomy is a curable and effective method. However, the recurrence rate is as high as 50%~70% in 5 years after surgery. Perioperative treatment with immunotherapy combined with target therapy is expected to improve the patient's prognosis. This study aims to evaluate the efficacy, safety and tolerability of camrelizumab combined with apatinib mesylate in the perioperative period of resectable hepatocellular carcinoma. The primary purpose of this study is to evaluate 2 year event-free survival（2y-EFS） of camrelizumab combined with apatinib mesylate in the perioperative period of hepatocellular carcinoma (CNLC Ib-IIIa). The secondary research purpose is to evaluate the R0 resection rate, the rate of subjects with major pathological response, the rate of subjects with pathological complete response, event-free survival (EFS) and overall survival of camrelizumab combined with apatinib mesylate in the perioperative period of resectable hepatocellular carcinoma. The safety and tolerability is also evaluated.

DETAILED DESCRIPTION:
Hepatocellular carcinoma (HCC) is the most common primary liver cancer. Hepatectomy is a curable and effective method. However, the recurrence rate is as high as 50%~70% in 5 years after surgery. Perioperative treatment with immunotherapy combined with target therapy is expected to improve the patient's prognosis. This study aims to evaluate the efficacy, safety and tolerability of camrelizumab combined with apatinib mesylate in the perioperative period of resectable hepatocellular carcinoma. This trial includes subjects with CNLC Ib/IIa/IIb/IIIa HCC. All eligible subjects will be randomized (1:1) to experimental group or control group. In the experimental group, patients will be treated with following: neoadjuvant therapy ( perioperative TACE treatment，camrelizumab and apatinib, 2 cycles), radical surgery, adjuvant therapy (camrelizumab and apatinib, 6 cycles); in the control group, patients will be treated with following: radical surgery,adjuvant therapy (camrelizumab and apatinib, 6 cycles). The primary purpose of this study is to evaluate 2 year event-free survival（2y-EFS） of camrelizumab combined with apatinib mesylate in the perioperative period of hepatocellular carcinoma (CNLC Ib-IIIa). The secondary research purpose is to evaluate the R0 resection rate, the rate of subjects with major pathological response, the rate of subjects with pathological complete response, event-free survival (EFS) and overall survival of camrelizumab combined with apatinib mesylate in the perioperative period of resectable hepatocellular carcinoma. The safety and tolerability is also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in this study and sign an informed consent form.
* Age ≥18 years old, no gender limit.
* Hepatocellular carcinoma confirmed by histopathology, cytology or imaging.
* CNLC stage Ib (single tumor with diameter ≥8 cm)/IIa/IIb/IIIa hepatocellular carcinoma, except for CNLC IIIa hepatocellular carcinoma combined with main portal vein tumor thrombus；multiple hepatocellular carcinoma was allowed to be treated with surgical excision combined with intraoperative ablation.
* Child-Pugh score: A grade (≤6 points).
* ECOG PS score: 0-1 points.

Exclusion Criteria:

* Known intrahepatic cholangiocarcinoma, sarcomatoid HCC, mixed cell carcinoma and fibrolamellar cell carcinoma; have other active malignancies other than HCC within 5 years or at the same time.
* Currently accompanied by interstitial pneumonia or interstitial lung disease.
* Existence of active autoimmune disease or history of autoimmune disease and may relapse.
* Patients with active infection, unexplained fever ≥38.5℃ within 1 week before randomization, or baseline white blood cell count >15*10^9/L.
* Patients with congenital or acquired immune deficiencies (such as HIV-infected persons).
* Those who are known to be allergic to any monoclonal antibodies, anti-angiogenesis targeted drugs or excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2023-01-31 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
2 year event-free survival（2y-EFS） | 2-year
  2y-EFS is defined as time from randomization to any of the following events: progression of disease that precludes surgery, local or distant recurrence, or death due to any cause.

SECONDARY OUTCOMES:
R0 resection rate | 30-day
  R0 resection rate
The rate of subjects of major pathological response (MPR) | 30-day
  MPR is defined as less than 10% residual tumor after neoadjuvant therapy of camrelizumab and apatinib therapy.
the rate of subjects with pathological complete response (pCR) | 30-day
  pCR is defined as no histologic evidence of malignancy or only the ingredients of carcinoma in situ was found in primary tumors.
Overall survival (OS) | 3-year
  OS is defined as the time from randomisation to death.
Event-free survival (EFS) | 3-year
  EFS is defined as the time from randomisation to tumor progression, postoperative relaspse or metastasis, or death, which occur first.
Disease-free survival (DFS) | 3-year
  DFS is defined as the time from randomization until disease recurrence or death from any cause.
Adverse event (AE) | 3-year
  Adverse events (AEs) ; serious adverse events (SAEs); surgery related safety.

CONTACTS AND LOCATIONS:
Overall Officials: Xuehao Wang, professor, Study Chair — The First Affiliated Hospital with Nanjing Medical University; Yongxiang Xia, Study Director — The First Affiliated Hospital with Nanjing Medical Univer
Locations (1):
- Jiangsu Province Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No